CLINICAL TRIAL: NCT05078255
Title: The Separate and Combined Effects of Long-term GIP and GLP-1 Receptor Activation in Patients with Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asger Lund, MD (Other)
Responsible Party: Sponsor-Investigator, Asger Lund, MD, Associate professor, MD PhD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1259-1491
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — semaglutide; Incretins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- placebo injections + placebo infusion (Placebo Comparator)
  Interventions: Other: Semaglutide 1.34 mg/ml placebo; Other: GIP placebo
- Semaglutide 1.34 mg/ml injections + GIP infusion (Experimental)
  Interventions: Drug: Semaglutide 1.34 MG/ML [Ozempic]; Drug: Glucose-dependent insulinotropic polypeptide (GIP)
- placebo injections + GIP infusion (Experimental)
  Interventions: Drug: Glucose-dependent insulinotropic polypeptide (GIP); Other: Semaglutide 1.34 mg/ml placebo
- Semaglutide 1.34 mg/ml injections + placebo infusion (Experimental)
  Interventions: Drug: Semaglutide 1.34 MG/ML [Ozempic]; Other: GIP placebo

INTERVENTIONS:
Drug: Semaglutide 1.34 MG/ML [Ozempic] — Semaglutide 1.34 mg/ml
  Other Names: Glucose-dependent insulinotropic polypeptide (GIP)
  Arms: Semaglutide 1.34 mg/ml injections + GIP infusion; Semaglutide 1.34 mg/ml injections + placebo infusion
Drug: Glucose-dependent insulinotropic polypeptide (GIP) — GIP
  Arms: Semaglutide 1.34 mg/ml injections + GIP infusion; placebo injections + GIP infusion
Other: Semaglutide 1.34 mg/ml placebo — Saline
  Arms: placebo injections + GIP infusion; placebo injections + placebo infusion
Other: GIP placebo — Saline
  Arms: Semaglutide 1.34 mg/ml injections + placebo infusion; placebo injections + placebo infusion

SUMMARY:
Due to reports of a severely reduced insulinotropic effect of the incretin hormone glucose-dependent insulinotropic polypeptide (GIP) in type 2 diabetes (T2D), GIP has not been considered therapeutically viable in T2D. Recently, however, tirzepatide, a novel dual incretin receptor agonist (activating both the GIP receptor and the glucagon-like peptide 1 (GLP-1) receptor) demonstrated massive improvements in glycaemic control and robust body weight losses; greater than observed with the GLP-1 receptor agonist semaglutide. However, the contribution of GIP receptor activation to these effects remains unknown. The present study will evaluate the glucose-lowering effect of GIP in the context of pharmacological GLP-1 receptor activation in patients with T2D.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
2. Men and women 18 to 74 years of age (both inclusive) at the time of signing informed consent
3. Diagnosed with type 2 diabetes for at least six months

   1. Treated with diet and exercise and/or stable metformin and/or sodium-glucose cotransporter 2 (SGLT-2) inhibitor and/or dipeptidyl-peptidase 4 inhibitor (DPP-4i) and/or sulfonylureas (SU) treatment for at least 3 months If treated with DPP-4i and/or SU, this treatment must be paused for 14 days prior to first CGM period in the trial
   2. HbA1c ≥48 to ≤91 mmol/mol
4. BMI ≥25 to ≤50 kg/m2
5. Stable body weight (less than 3 kg self-reported change during the previous 90 days)

Exclusion Criteria:

For an eligible participant, all exclusion criteria must be answered "no".

1. Diagnosed with type 1 diabetes
2. Known or suspected hypersensitivity to trial product or related products
3. Acute decompensation of glycaemic control requiring immediate intensification of treatment to prevent acute complications of diabetes (e.g. diabetes ketoacidosis) which required help from doctor or hospitalisation within 90 days prior to screening
4. Previous participation in this trial. Participation is defined as signed informed consent. Participation is allowed if the protocol is updated to a newer version
5. Participation in another clinical trial within 90 days before screening
6. Woman who are pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods (intrauterine devices or hormonal contraception (oral contraceptive pills, implants, transdermal patches, vaginal rings or long-acting injections))
7. If previously treated with GLP-1RA, information about the time and reason for stopping will be collected. Based upon this, the eligibility will be judged by the investigator
8. Participation in an organised weight reduction programme within 3 months before screening
9. Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol
10. Anticipated change in lifestyle (e.g. smoking, eating or exercise pattern) during the trial
11. Any laboratory safety parameter at screening outside the below extended laboratory ranges, see laboratory manual for specific values

    * Albumin outside lower normal limit (LNL) -5% and upper normal limit (UNL) +5%
    * Alanine aminotransferase (ALT) outside LNL -100% and UNL +50%
    * Creatinine outside UNL +10%
    * Haemoglobin outside LNL -5% and UNL +10%
    * Leukocytes outside LNL -20% and UNL +20%
    * Thrombocytes outside LNL -15% and UNL +15%
    * Bilirubin (total) outside UNL +15%
    * Amylase ≥ UNL +100%
12. Untreated or uncontrolled hypothyroidism/hyperthyroidism defined as thyroid-stimulating hormone (TSH) <0.4 mIU/L or > 6 mIU/L
13. Obesity related to endocrinologic disorders (e.g. Cushing Syndrome)
14. Any blood draw in excess of 25 mL in the past month, or donation of blood or plasma in excess of 400 mL within the 90 days preceding screening
15. Use of any prescription or non-prescription medication (apart from oral contraceptives, routine vitamins, occasional use of paracetamol, acetylsalicylic acid, or ibuprofen) which could interfere with pharmacokinetic or pharmacodynamic results, as judged by the investigator, such as:

    * herbal products and non-routine vitamins
    * Glucose lowering medication (except metformin)
    * medication that may cause weight gain, including systemic corticosteroids, tricyclic antidepressants, and atypical antipsychotics
    * orlistat, zonisamide, topiramate, phentermine, lorcaserin, bupropion, naltrexone or other weight loss drugs
    * Blood pressure and lipid lowering agents (e.g. statins) drugs are allowed if treatment has been stable for ≥ 1 month prior to screening and treatment should preferably be kept unchanged during the trial
16. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
17. History of pancreatitis (acute or chronic)
18. History of major depressive disorder or other severe psychiatric disorders, e.g. schizophrenia or bipolar disorder within the last 2 years or lifetime history of suicide attempt
19. Surgery scheduled for the trial duration period, except for minor, non-gastrointestinal surgical procedures at the discretion of the investigator
20. Sitting blood pressure (after resting for at least 5 minutes) ≥160 mmHg systolic or ≥ 100 mmHg diastolic or heart rate of ≥ 90 beats/min after resting for at least 5 minutes (if white-coat hypertension is suspected, one repeat measurement is allowed; last measure being conclusive and to be recorded in the case report form (CRF))
21. Cancer (past or present, except basal cell skin cancer or squamous cell skin cancer), which in the investigator's opinion could interfere with the results of the trial
22. Known or suspected alcohol abuse within 1 year from screening (defined as regular intake of more than 14 units weekly for men and 7 units weekly for women - one unit of alcohol equals about 300 mL of beer or lager, one glass (100 ml) of wine, or 25 ml spirits) or a positive result of an alcohol test
23. Known or suspected drug/chemical substance abuse within 1 year from screening
24. Inability or unwillingness to perform self-injection at the screening visit (with a placebo test pen)
25. Mental incapacity, language barriers or unwillingness to comply with the requirements of the protocol, which may preclude adequate understanding or co-operation during the trial, as judged by the investigator
26. Investigator, any sub-investigators, research assistants, pharmacist, trial coordinators, other staff, sponsor staff or relatives thereof directly or indirectly involved in the conduct of the trial cannot participate in the trial

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Mean glucose levels (assessed by blinded continuous glucose monitoring (CGM)) | 14-day mean glucose levels during the last 14 days of the intervention period as compared to 14-day mean glucose levels during the last 14 days of the run-in period.
  The primary outcome is change in 14-day mean glucose levels (assessed by CGM) during the last 14 days of the intervention period as compared to 14-day mean glucose levels during the last 14 days of the run-in period.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Capital Region, Denmark

REFERENCES:
- [Derived] Helsted MM, Gasbjerg LS, Vilsboll T, Nielsen CK, Forman JL, Christensen MB, Knop FK. Separate and combined effects of long-term GIP and GLP-1 receptor activation in patients with type 2 diabetes: a structured summary of a study protocol for a double-blind, randomised, placebo-controlled clinical trial. BMJ Open. 2023 Feb 27;13(2):e065736. doi: 10.1136/bmjopen-2022-065736. PMID 36849212